CLINICAL TRIAL: NCT00201760
Title: A Randomized Phase II Study of Gemcitabine/ Trastuzumab and Gemcitabine/ Cisplatin/ Trastuzumab in Patients With Metastatic Breast Cancer
Brief Title: Gemcitabine/ Trastuzumab and Gemcitabine/ Cisplatin/ Trastuzumab in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kari Kendra (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Kari Kendra, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0342
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; Trastuzumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 Gemcitabine/Cisplatin/Trastuzumab (Experimental): Gemcitabine 1000 mg/m2 iv over 30 minutes on days 1 and 8 Cisplatin 30 mg/m2 iv over 90 minutes on days 1 and 8 Trastuzumab 2 mg/kg iv over 30 minutes on days 1, 8 and 15 (if trastuzumab was not administered within the past 3 weeks, a loading dose of 4 mg/kg iv over 90 minutes will be given on the first day of cycle 1 only).
  Interventions: Drug: Gemcitabine; Drug: Trastuzumab; Drug: Cisplatin
- Arm 2 Gemcitabine / Trastuzumab (Active Comparator): Gemcitabine 1000 mg/m2 iv over 30 minutes on days 1 and 8 Trastuzumab 2 mg/kg iv over 30 minutes on days 1, 8 and 15 (if trastuzumab was not administered within the past 3 weeks, a loading dose of 4 mg/kg iv over 90 minutes will be given on the first day of cycle 1 only).
  Interventions: Drug: Gemcitabine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 IV over 30 minutes on Days 1 and 8.
  Other Names: Gemzar
Drug: Trastuzumab — 2 mg/kg IV on days 1, 8 and 15. If Trastuzumab has not been administered within the 3 weeks before starting this treatment, the first dose of Trastuzumab given on Cycle 1, Day 1 will be 4 mg/kg followed by 2 mg/kg weekly.
  Other Names: Herceptin
Drug: Cisplatin — 30 mg/m2 IV on Day 1 and Day 8.
  Other Names: Platinol®-AQ; CDDP
  Arms: Arm 1 Gemcitabine/Cisplatin/Trastuzumab

SUMMARY:
This study determines the proportion of metastatic breast cancer patients progression free after 6 months when treated with gemcitabine/ cisplatin/ trastuzumab or gemcitabine/ trastuzumab.

DETAILED DESCRIPTION:
Rationale: Previous studies have demonstrated the anti-tumor efficacy of gemcitabine and trastuzumab against metastatic breast cancer when given alone and in combination. Yet, research indicates that the two drugs given together work more effectively than either alone. Laboratory studies testing the combination of trastuzumab and cisplatin have shown synergistic anti-tumor activity with the two drugs. In addition, clinical studies suggest a high level of anti-tumor activity with the combination of gemcitabine and cisplatin. Researchers are testing the triple drug combination of gemcitabine, trastuzumab, and cisplatin in the current study to evaluate the potential for enhanced responsiveness in patients with Her-2/neu overexpressing breast cancer as well as comparing it to the double drug combination of gemcitabine and trastuzumab.

Purpose: This study will measure patient responses and compare the efficacy of a double drug combination (gemcitabine and trastuzumab) with a triple drug combination (gemcitabine, trastuzumab, and cisplatin) in patients with metastatic breast cancer. Side effects will be carefully assessed in patients.

Treatment: Patients in this study will receive one of two treatment combinations. A computer will randomly assign patients to a treatment group. Group one will be given gemcitabine and trastuzumab. Gemcitabine will be given to patients on days 1 and 8, and trastuzumab on days 1, 8, and 15. Group two will receive gemcitabine, trastuzumab, and cisplatin. Gemcitabine and cisplatin will both be administered on days 1 and 8, and trastuzumab on days 1, 8, and 15. Each treatment cycle (for both groups) will last a total of 21 days. All study drugs will be administered through intravenous infusions. Several tests and exams will be given throughout the study to closely monitor patients. Thorough patient exams will be given at the beginning of each treatment cycle. Imaging tests will be done every two cycles for the first eight cycles and then every three cycles until study completion. Study treatment will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Eligibility Criteria:

* Must have invasive metastatic breast cancer
* Tumor must be Her 2/neu 3+ by IHC (must be confirmed by Ohio State University pathology)or positive FISH
* Histological confirmation of invasive breast cancer either from the original diagnosis and/or diagnosis of metastatic disease.
* Tumor must be detectable clinically or radiographically (a positive bone scan is allowed as the only site of disease). Unidimensional measurements must be obtained whenever possible). Bone marrow only disease is not eligible for enrollment on this study.
* No evidence of congestive heart failure, symptoms of coronary artery disease, serious cardiac arrhythmias, or evidence of prior myocardial infarction on EKG or ECHO. Patients must have normal LV function and LVEF(left ventricular ejection fraction)> 50% as demonstrated by either echo or muga within the proceeding 4 weeks.
* Must have adequate renal and hepatic function documented by a serum creatinine < 1.5 x the institutional upper limit of normal (ULN), serum bilirubin <1.5 x ULN and liver enzymes (AST, ALT, or alkaline phosphatase) < 2 x ULN (< 5 x ULN if hepatic metastasis) within 21 days prior to registration.
* Patients must have an ANC (absolute neutrophil count) > 1.5, platelets > 100,000, Hemoglobin >9.0 within 21 days of registration.
* If patients are on bisphosphonates at the time of registration, with a stable creatinine over the preceding 2 months, then they may continue bisphosphonates during the study.
* No more than one prior Trastuzumab/chemotherapy or Trastuzumab/biotherapy combination for metastatic disease. Additional Trastuzumab therapy may have been given in the adjuvant setting. Prior hormonal therapy is allowed for either adjuvant or metastatic disease.
* Must be >3 weeks since administration of last chemotherapy prior to initiation of treatment on this trial. Prior trastuzumab may have been administered within one week of initiation of treatment on this trial if the last dose was 2 mg/kg. Any prior trastuzumab dosing greater than 2 mg/kg requires a 3 week washout period.
* Patients may have received prior cisplatin or carboplatin for metastatic disease.
* No CNS(central nervous system)metastasis disease.
* No active infection at time of registration.
* Pregnant or nursing women may not participate in trial.
* Patients must be informed of the investigational nature of this study and sign and give written informed consent in accordance with institutional and federal guidelines.
* ECOG (Eastern Cooperative Oncology Group)performance status < 2 at the time of registration.
* Patients may participate in a non-treatment related protocol while participating in this study.
* No other active malignancy is allowed. Adequately treated basal cell, squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-02-25 (Actual); Primary Completion 2009-10-31 (Actual); Study Completion 2009-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Kendra, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Egger SJ, Chan MMK, Luo Q, Wilcken N. Platinum-containing regimens for triple-negative metastatic breast cancer. Cochrane Database Syst Rev. 2020 Oct 21;10(10):CD013750. doi: 10.1002/14651858.CD013750. PMID 33084020
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in the study from February 2005 to March 2008
Period: Overall Study
Arm/Group | Arm 1 Gemcitabine/Cisplatin/Trastuzumab | Arm 2 Gemcitabine / Trastuzumab
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Gemcitabine/Cisplatin/Trastuzumab | Arm 2 Gemcitabine / Trastuzumab | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Full Range); unit: years] | 51 [33 to 62] | 42 [36 to 57] | 47.5 [33 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression
Description: Proportion of patients with metastatic breast cancer free of disease progression at 6 months following treatment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Gemcitabine/Cisplatin/Trastuzumab | Arm 2 Gemcitabine / Trastuzumab
Number analyzed (Participants) | 5 | 5
Participants | 1 | 0

2. Secondary Outcome: Measure Response Rate of Each Drug Combination
Description: Response rate of the of the triple drug combination therapy and the double drug combination therapy regimens.
Time Frame: Up to 24 months
Measure: Number; unit: patients
Arm/Group | Arm 1 Gemcitabine/Cisplatin/Trastuzumab | Arm 2 Gemcitabine / Trastuzumab
Number analyzed (Participants) | 5 | 5
patients | 1 | 0

3. Secondary Outcome: Number of Participants With Grades 3 and Grade 4 Toxicity Profiles of the Drug Combinations
Description: Adverse Events will be graded in accordance with the CTCAE Version 3.0 Toxicity grading criteria
Time Frame: Up to 24 months
Population: Grades 3 and Grade 4
Measure: Number; unit: patients
Arm/Group | Arm 1 Gemcitabine/Cisplatin/Trastuzumab | Arm 2 Gemcitabine / Trastuzumab
Number analyzed (Participants) | 5 | 5
patients
  Leukocytes (total WBC) | 2 | 1
  Neutrophils/granulocytes | 2 | 2
  Platelets (Thrombocytopenia) | 1 | 0
  Fatigue | 1 | 1

ADVERSE EVENTS:
Description: Adverse Events were graded in accordance with the NCI CTC Version 3.0 Toxicity grading criteria.
Arm/Group | Arm 1 Gemcitabine/Cisplatin/Trastuzumab | Arm 2 Gemcitabine / Trastuzumab
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Gemcitabine/Cisplatin/Trastuzumab (N=5) | Arm 2 Gemcitabine / Trastuzumab (N=5)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Nausea/vomiting/diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Gemcitabine/Cisplatin/Trastuzumab (N=5) | Arm 2 Gemcitabine / Trastuzumab (N=5)
Hemoglobin (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Leukocytes (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Neutrophils (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 4 (4)
Fever (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4)
Weight loss (Investigations) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hot Flashes (Vascular disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Elevated ALT (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Elevated AST (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Mood alteration (depression) (Psychiatric disorders) | 2 (2) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes